CLINICAL TRIAL: NCT00752661
Title: An Exploratory Study of an Active Ingredient of JNS013-tramadol Hydrochloride in Patients With Osteoarthritis of the Knee or Low Back Pain
Brief Title: An Exploratory Study of Tramadol Hydrochloride in Patients With Osteoarthritis of the Knee or Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013900
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-08

CONDITIONS: Osteoarthritis; Low Back Pain
Keywords: osteoarthritis; low back pain; oral drug; tramadol
MeSH Terms: conditions — Osteoarthritis; Low Back Pain | interventions — Tramadol

INTERVENTIONS:
Drug: Tramadol Hydrochloride; JNS013

SUMMARY:
The purpose of this study is to find the clinical dose range of an active ingredient of JNS013 - Tramadol hydrochloride in chronic-pain patients who cannot attain a sufficient analgesic effect from non-steroidal anti-inflammatory drugs (NSAIDs).

DETAILED DESCRIPTION:
Since JNS013 is a combination of tramadol hydrochloride (TRAM) acting as a weak opioid with acetaminophen (APAP) inhibiting central COX-3, it is expected to have an intermediate effect between narcotic analgesics and NSAIDs (non-steroid anti-inflammatory drugs). This is a multicenter, open-label, dose response study. The purpose of this study is to find the clinical dose range of TRAM in patients with chronic pain due to osteoarthritis (OA) of the knee or low back pain (LBP) who cannot attain a sufficient analgesic effect from NSAIDs. The investigational product will be orally administered 4 times daily (after each meal and before bedtime) at a dose of 25 to 100 mg at least 4-hour intervals. Treatment will be started at an initial dose of 100 mg/day, and the dose is titrated by 25 mg every 7 days if the analgesic effect is insufficient and there is no problem with the safety. Treatment will be continued up to 35 days in total at a dose of 400 mg/day or a dose of which a sufficient analgesic effect can be obtained. The primary efficacy endpoint is the change in the intensity of pain from the beginning of dose-finding period (baseline) to the final assessment point (Up to Day 36), by using VAS (Visual Analog Scale). The safety evaluations are adverse events, laboratory examinations, blood pressure/pulse rate and body weight. Total study period of this study is 49days, Screening period is 7days, Administration period is 35 days and Follow-up period is 7 days. The investigational product will be orally administered 4 times daily (after each meal and before bedtime) at a dose of 25 to 100 mg at least 4-hour intervals. Treatment will be started at an initial dose of 100 mg/day, and the dose is titrated by 25 mg every 7 days if the analgesic effect is insufficient and there is no problem with the safety. Treatment will be continued up to 35 days in total at a dose of 400 mg/day or a dose of which a sufficient analgesic effect can be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain due to OA of the knee or LBP that persists for more than 3 months at the initiation of the observation period
* Patients who received oral NSAIDs at a usual highest dose for at least 14 consecutive days during 3 months before the initiation of the observation period, but could not attain a sufficient analgesic effect
* Patients with the intensity of the strongest pain during 48 hours before the initiation of the observation period is >= 40 mm and < 80 mm on VAS
* Ambulatory outpatients
* Prior to the conduct of the study, patients who were given a sufficient explanation about the investigational product and this study and have given their own consent in writing to participate in the study.

Exclusion Criteria:

* Patients with conditions for which opioids are contraindicated
* Patients with a hypersensitivity to opioids
* Patients who received TRAM in the past and discontinued the treatment due to ineffectiveness or adverse reactions
* Patients with complications associated with pain to the degree considered to have an influence on the efficacy assessment (trauma such as fracture, headache, post-herpetic neuralgia)
* Patients with a complication of severe spinal disease

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change in the intensity of pain from the beginning of dose-finding period (baseline) to the final assessment point, by using VAS.

SECONDARY OUTCOMES:
Percentage of patients considered analgesic effect present based on the change in VAS, VAS on each assessment day, PI (pain intensity rating), PAR (pain relief rating), PID (pain intensity difference), PRID (pain relief combined with pain intensity).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.

REFERENCES:
- See also: An exploratory study of an active ingredient of JNS013 - tramadol hydrochloride in patients with osteoarthritis of the knee or low back pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=414&filename=CR013900_CSR.pdf